CLINICAL TRIAL: NCT02941783
Title: Drug Use Investigation of Kovaltry in Hemophilia A Patients
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18706; 2015/01011 (Other: Company Internal)
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Hemophilia A
Keywords: Kovaltry; hemophilia A; Japan; Post-marketing surveillance
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human; Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BAY81-8973: Hemophilia A patients who require Factor VIII replacement therapy
  Interventions: Drug: Kovaltry (Antihemophilic Factor [Recombinant], BAY81-8973)

INTERVENTIONS:
Drug: Kovaltry (Antihemophilic Factor [Recombinant], BAY81-8973) — Treatment parameters following the physician's decision based on the summary of product characteristics.

SUMMARY:
The objective in this study is collecting post-marketing information on the safety and efficacy of Kovaltry under the routine clinical practice.

DETAILED DESCRIPTION:
This company-sponsored study is a single-arm, prospective, observational study in hemophilia A patients administered Kovaltry. 200 cases will be planned to be registered as safety analysis set in three-year period. Within 200 cases, 50 cases less than 12 years old will be planned to be registered. Target population are all hemophilia A patients. The treatment should be performed based on the product label in Japan. The standard observation period is two years.

ELIGIBILITY:
Inclusion Criteria:

* Male and female hemophilia A patients.
* Patients for whom the decision to treat with Kovaltry was determined prior to enrollment in the study.

Exclusion Criteria:

* Patients participating in an investigational program with interventions outside of routine clinical practice.
* Patients with an additional diagnosis of any bleeding/coagulation disorder other than hemophilia A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female hemophilia A patients are registered after the decision for treatment with Kovaltry has been made by the investigator. Both 'on demand' and 'prophylaxis' treatment are included.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as measure of safety and tolerability | Up to 2 years
Number of participants with serious adverse events as measure of safety and tolerability | Up to 2 years

SECONDARY OUTCOMES:
Number of annual bleeds | Up to 2 years
Efficacy of controlling of bleeds | Up to 2 years
  The efficacy is evaluated by the investigator and given on a four point scale: Excellent, Good, Moderate and Poor.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Multiple Locations, Japan